CLINICAL TRIAL: NCT05312424
Title: Effect of Annatto-derived Geranylgeraniol (GG) on Statin-associated Myopathy
Brief Title: Annatto-derived GG for Statin-associated Myopathy
Acronym: GG-statin
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: L22-130
Record Dates: First submitted 2022-03-09; First posted 2022-04-05 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Myopathy; Primary
MeSH Terms: conditions — Muscular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo group: subject will take one pill (150 mg olive oil) after breakfast and another pill (150 mg olive oil) after dinner
  Interventions: Dietary Supplement: Placebo
- Low GG (Active Comparator): LOW GG group: subject will take one pill (150 mg olive oil) after breakfast and another pill (150 mg GG) after dinner
  Interventions: Dietary Supplement: Low GG
- High GG (Active Comparator): HIGH GG group: subject will take one pill (150 mg GG) after breakfast and another pill (150 mg GG) after dinner
  Interventions: Dietary Supplement: High GG

INTERVENTIONS:
Dietary Supplement: Placebo — 300 mg olive oil
  Arms: Placebo
Dietary Supplement: Low GG — 150 mg GG
  Arms: Low GG
Dietary Supplement: High GG — 300 mg GG
  Arms: High GG

SUMMARY:
To evaluate the effects of 3-months annatto-derived geranylgeraniol (GG) supplementation on statin-associated skeletal muscle health.

DETAILED DESCRIPTION:
Statins are widely prescribed cholesterol-lowering oral drugs. The majority of reported adverse effects due to statin include muscle pain, weakness, cramp, and tiredness. CoQ10 supplementation has been widely used to reduce statin-related muscle complaints. Several human studies have been reported with inconsistent effects of CoQ10 on statin-related symptoms. This study is to investigate the role of 3-month annatto-derived geranylgeraniol (GG) in statin-related muscle outcomes in humans. Qualified subjects will be matched by age, gender, and body weight, and then randomly assigned to a no GG group, a low GG dose group, or a high GG dose group. The outcome measures will be assessed at baseline and after 3 months. Muscle-associated measurements will be recorded using subject questionnaires (also follow-up after 3 and 6 months), muscle performance results, and blood samples. We will monitor the safety of subjects after 3 months. Food intake, physical activity, and medication changes will be recorded at baseline and after 3 months. All data will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥40 of either sex
* Statin-treated patients with muscle pain alone or accompanied by other symptoms.
* Patients currently receiving a statin who developed new-onset myalgias in within 90 day of initiation or a dosage increase

Exclusion Criteria:

* Malignancy or significant neurological or psychiatric disturbances, including alcohol or drug abuse.
* Woman who is pregnant, breastfeeding, or of childbearing potential and not taking adequate contraceptive precautions.
* Had CoQ10 supplement one month before starting the study.
* Genetic musculoskeletal and neurologic disorder known to affect skeletal muscle metabolism
* Had steroid medication one month before starting the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
SAMS-CI | change in SAMS-CI at 3 months
  Statin-Associated Muscle Symptom Clinical Index (SAMS-CI) is to assess muscle pain, muscle weakness, tiredness, and cramps.
BPI | change in BPI at 3 months
  Brief Pain Inventory (BPI) is to assess pain and interference of pain with everyday life.

SECONDARY OUTCOMES:
Lower body isometric strength | change in lower body isometric strength at 3 months
  Lower body (i.e., predominantly of the quadriceps and hip extensors) isometric strength is measured using a dynamometer
Functional lower body strength | change in functional lower body strength at 3 months
  Functional lower body strength is measured using a loaded 50m walk.
Wall-sit test | change in wall-sit test at 3 months
  Wall-sit test (wall-slide test) is to assess static leg strength and endurance, particularly of the quadriceps and hip extensors
Heel raise test | change in heel raise test at 3 months
  Heel raise test is commonly used to test calf muscle endurance, function, and performance. Single-leg or both-leg raise will be tested while staining on a step bench
blood biomarkers: serum creatinine kinase activity | change in serum creatinine kinase activity at 3 months
  Creatine kinase is to assess muscle damage.
blood biomarkers: myostatin | changes in serum myostatin at 3 months
  Myostatin is to assess muscle damage
blood biomarkers: atrogin 1 | changes in serum atrogin 1 at 3 months
  atrogin 1 is to assess muscle damage
blood biomarkers: hsCRP | changes in serum hsCRP at 3 months
  hsCRP is to assess inflammation
blood biomarker: IL-6 | changes in serum IL-6 at 3 months
  IL-6 is to assess inflammation
blood lipid profiles | changes in blood lipid profiles at 3 months
  lipid profiles include total triglycerides, total cholesterol, HDL, and calculated LDL
plasma menaquinone-4 (MK4) + menaquinone-4 (MK7) | changes in plasma MK4+MK7 at 3 months
  MK4 and MK4 are vitamin K2 homologues and are measured by HPLC

CONTACTS AND LOCATIONS:
Overall Officials: Chwan-Li (Leslie) Shen, PhD, Principal Investigator — Texas Tech Health Science Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No